CLINICAL TRIAL: NCT03322943
Title: The Comparison About the Response of Ursodeoxycholic Acid in Primary Biliary Cholangitis Only and Primary Biliary Cholangitis With High Immune Globulin G or Aminotransferase at West China Hospital
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Li Yang, Principal Investigator, West China Hospital
Other Study IDs: PBC-2
Record Dates: First submitted 2017-10-08; First posted 2017-10-26 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Primary Biliary Cholangitis
Keywords: Ursodeoxycholic Acid; Response
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the different response of Ursodeoxycholic Acid in primary biliary cholangitis only and primary biliary cholangitis with high immune globulin G or aminotransferase at West China Hospital from 2008-2017.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with primary biliary cholangitis Treated with Ursodeoxycholic Acid in West China Hospital for at least 1 year

Exclusion Criteria:

Autoimmune hepatitis Primary sclerosing cholangitis

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with primary biliary cholangitis and treated with Ursodeoxycholic Acid at West China Hospital by review of medical records.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Description of demographics, clinical index after treatment | up to 1 year
  age，sex，ALT（IU/L），AST（IU/L），ALP（IU/L），GGT（IU/L）,IgG（g/L）

SECONDARY OUTCOMES:
Evaluation whether the PBC patients have response after treatment | within 1 year
  Use Paris II criterion to estimate

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, MD, Study Chair — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China